CLINICAL TRIAL: NCT04067557
Title: Diagnosis of Bacterial Vaginosis Using Molecular PCR Test.
Brief Title: Diagnosis of Bacterial Vaginosis Comparing Modified Hay/Ison With Molecular Diagnosis
Status: Completed | Type: Observational
Sponsor: Skaraborg Hospital (Other Government)
Responsible Party: Principal Investigator, Per-Goran Larsson, professor, Skaraborg Hospital
Other Study IDs: BV
Record Dates: First submitted 2019-08-19; First posted 2019-08-26 (Actual); Last update posted 2019-08-28 (Actual); Status verified 2019-08

CONDITIONS: Infection, Bacterial
MeSH Terms: conditions — Bacterial Infections

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — PCR diagnosis
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: molecuar test of BV — diagnosis of BV

SUMMARY:
Among 300 women that are scheduled a therapeutic abortion screening diagnopsis of BV are done using Gram stained vaginal smear and with a molecular test using PCR for 5 different bacteria.

DETAILED DESCRIPTION:
The molecular test will test for Atophobium vaginae, Leopitrichia spp, Megasphaera Mobiluncus and BVAB2

ELIGIBILITY:
Inclusion Criteria:

women scheduled a therapeutic abortion (Before 12th week) will be screened for gential infections such as chlamydia and Gc together with bacterial vaginosis

Exclusion Criteria:

* women not pregnat

Age Groups: Child, Adult, Older Adult
Study Population: women that are scheduled a therapeutic abortion screening visiting Skaraborg hospital Sweden
Sampling Method: Non-Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2013-01-01 (Actual); Primary Completion 2013-05-01 (Actual); Study Completion 2013-06-01 (Actual)

PRIMARY OUTCOMES:
Diagnosis of bacterial vaginosis comparing modified Hay/Ison with molecular diagnosis | 4 month
  Comparing the Gram stained vaginal smears using Hay/Ison (i.e. BV or normal) criteria with a molecular PCR method with 5 different bacterium and after an algoritm end up with the result (i.e. BV or normal). The number of women with the diagnosis of BV with each of the diagnostic test can be compared calculatitng a KAPPA index

CONTACTS AND LOCATIONS:
Overall Officials: P-G Larsson, Principal Investigator — professor
Locations (1):
- Department of Ob/Gyn, Skaraborgshospital Skövde, Skövde, Sweden